CLINICAL TRIAL: NCT01573364
Title: Evaluation of the Prevalence and the Reversibility of the Lung Hyperinflation in Uncontrolled Persistent Asthmatic Patients With Dyspnea
Brief Title: Prevalence and Reversibility of Lung Hyperinflation in Asthma
Acronym: Dist'air2
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: EQFST5213
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Asthma
Keywords: Distal Airways; Hyperinflation; Reversibility
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this observational study is to evaluate the pulmonary hyperinflation and its immediate reversibility to a short acting beta2 agonist test in uncontrolled persistent asthmatic patients with dyspnea.

DETAILED DESCRIPTION:
The other objectives are :

* the evaluation of the hyperinflation defined by an increase of the residual volume (RV),
* the observation of the relationship between the hyperinflation and the asthma characteristics,
* the study of the improvement of the functional parameters after a reversibility test
* the evaluation of the correlation between hyperinflation parameters evolution, chest tightness and dyspnea

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of uncontrolled persistent asthma (ACT </= 19) or with an MRC score of dyspnea >/= 1
* Patient requiring a check-up including a pulmonary function test by plethysmography with a reversibility test

Exclusion Criteria:

* Patient participating to an other clinical trial or having participated to a clinical trial with medicine in the last 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Capucine de Meynard, MD, Study Director — Chiesi S.A.; Daniel Dusser, MD, Prof, Study Chair — Hopital Cochin Paris France
Locations (1):
- Laboratoire Chiesi S.A., Courbevoie, France

REFERENCES:
- [Derived] Perez T, Chanez P, Dusser D, Devillier P. Prevalence and reversibility of lung hyperinflation in adult asthmatics with poorly controlled disease or significant dyspnea. Allergy. 2016 Jan;71(1):108-14. doi: 10.1111/all.12789. Epub 2015 Nov 6. PMID 26466328